CLINICAL TRIAL: NCT06798636
Title: Investigating the Effects of a Psychedelic-augmented Mental Imagery-based Intervention for Young People With Self-harm Behaviour: an Experimental Medicine Study
Brief Title: PsiloIMAGINE: A Psychedelic-augmented Mental Imagery-based Intervention for Young People With Self-harm
Acronym: PsiloIMAGINE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 172441; IRAS ID: 330839 (Other: Health Research Authority)
Record Dates: First submitted 2025-01-14; First posted 2025-01-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Self Harm
Keywords: Psilocybin; Psychedelic; Self injury; Self-Injurious Behaviour
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin 5mg (Experimental): Participants will be given orally one 5mg psilocybin capsule.
  Interventions: Drug: Psilocybin 5 mg with cognitive behavioural therapy intervention
- Placebo (Placebo Comparator): Participants will be given orally one 25mg MCC inert placebo capsule.
  Interventions: Drug: Placebo with cognitive behavioural therapy intervention

INTERVENTIONS:
Drug: Psilocybin 5 mg with cognitive behavioural therapy intervention — This is an oral 5mg psilocybin dose preceding a mental imagery rescripting procedure
  Other Names: Psilocybin
  Arms: Psilocybin 5mg
Drug: Placebo with cognitive behavioural therapy intervention — This is an oral placebo comparator preceding a mental imagery rescripting procedure
  Arms: Placebo

SUMMARY:
Approximately 20% of young people experience self-harm behaviour in their lives. Self-harm can occur across different mental health disorders, and lead to negative outcomes and risk of suicide. Current treatments are long, costly and do not suit all young people, making it essential to research alternative treatments. Therapy combined with psychedelic drugs has recently been shown to be helpful in a variety of mental health disorders, including depression. This research project will explore the mechanisms by which combining a low dose of psychedelic psilocybin with a cognitive technique may target self-harm behaviour in young people (aged 16-25).

Previous research has shown that mental images of self-harm are common among individuals who self-harm and can increase the urge to self-harm. Imagery Re-Scripting (ImRS) is a cognitive technique that guides an individual to replace mental imagery driving self-harm with an alternative image that will instead discourage self-harm and promote alternative coping strategies. However, during ImRS individuals may fear bringing negative mental images and emotions to mind, hindering the process. Psychedelic substances can increase the ability to tolerate difficult emotions, make thinking styles more flexible and individuals more open to change. Based on this, the aim is to test if enhancing a cognitive technique with a low dose psychedelic can modify the cognitive mechanisms maintaining self- harm behaviour.

The aim is to examine the effect of a sub-hallucinogenic dose of psilocybin in combination with ImRS on cognitive processes, such as experiencing vivid mental images, and whether it can reduce these mental images and associated negative emotions in young people with recent self-harm behaviour above the effects of ImRS alone.

The hypothesis is that psilocybin could facilitate confronting the emotions that arise during ImRS and make it easier to generate new helpful mental imagery.

These experimental data could lay the foundation for future treatment development targeting self-harm in young people.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 lifetime episodes of self-harm measured using the Self-Injurious Thoughts and Behaviours Interview (Nock et al., 2007) and at least 1 self-harm episode in the past month
* Self-harm-associated mental imagery in the past 6-weeks measured using the Self-harm Imagery Interview (Hales et al., 2011)
* Any gender
* Age: 16-25 years old
* Good command of the English language
* Mental capacity to provide written informed consent
* Participant is willing to engage in tasks showing images of self-harm
* Participant is willing to talk about mental health and self-harm behaviour
* Normal ECG and blood pressure (determined by study medic)
* Psychedelic naïve
* No recreational drug use 7 days prior to the dosing visit
* Comfortable using a computer and smartphone app for data collection, access to the internet from home and willing to have some of the study visits via video-link

Exclusion Criteria:

* Current or past history of psychosis or mania in themselves or a first-degree relative
* Current severe suicidal ideation that constitutes a risk for their participation
* Have a medically significant condition which renders them unsuitable for the psychedelic component of the study (e.g., hypertension, diabetes, severe cardiovascular disease, hepatic or renal failure etc.)
* Previous psychedelic use
* Current or chronic history of kidney or liver disease
* Have previously experienced a serious adverse response after psychedelic use
* Intoxication on any of the visits, as assessed by difficulty in walking, the slurring of speech, difficulty concentrating or drowsiness
* Clinically significant head injury (e.g., requiring medical or surgical intervention) that in the opinion of the investigators, contraindicates their participation
* Severe learning disability (including dyslexia/dyspraxia) that needs support to perform daily work/school tasks
* Unwillingness or inability to follow the procedures outlined in the protocol
* Are currently using a psychoactive medication
* History of psychosurgery
* In the opinion of the study team, they are unlikely to comply with the study protocol and lifestyle restrictions that it imposes
* Unstable physical illness
* Heavy smoker
* Those needing regular specified medication that might interact adversely with psilocybin e.g., selective serotonin reuptake inhibitor, 5HT1 agonists, mirtazapine, trazodone, analgesics that have serotonergic effects (tramadol), MAOI's, antipsychotics with significant 5-HT2A receptor antagonist actions (risperidone, olanzapine, and quetiapine)
* Those unwilling to allow their GP or involved mental health practitioners to be informed of their participation
* Women of childbearing age who are not using reliable contraceptive methods
* Women of childbearing age who are unable to comply with or produce a positive pregnancy urine test

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of mental imagery | Up to 3 months
  Frequency scores on a 1-10 Likert scale related to self-harm and novel adaptive mental imagery
Vividness of mental imagery | Up to 3 months
  Vividness scores on a 1-10 Likert scale related to self-harm and novel adaptive mental imagery
Intensity of emotions related to mental imagery | Up to 3 months
  Emotions' intensity scores on a 1-10 Likert scale related to self-harm and novel adaptive mental imagery
Believability of cognitions related to mental imagery | Up to 3 months
  Cognitions' believability scores on a 1-10 Likert scale related to self-harm and novel adaptive mental imagery
Schemas | Up to 3 months
  Scores on Young Schema Questionnaire Short Form (Young et al., 1994)

SECONDARY OUTCOMES:
Approach Avoidance task | Up to 5 months
  Performance (e.g., reaction time, accuracy) to self-harm vs neutral pictures and positive vs neutral pictures on the Approach Avoidance task (Loijen et al., 2020)
Probabilistic Reversal Learning Task | Up to 5 months
  Performance (e.g., reaction time, accuracy, learning rate) on the Probabilistic Reversal Learning task (Dombrovski et al., 2010)
Self-harm Dot Probe Task | Up to 5 months
  Performance (e.g., reaction time, accuracy, learning rate) on the Self-harm Dot Probe Task (Constantinou et al., 2010)
Difficulty in Emotional Regulation | Up to 5 months
  Scores on the Difficulty in Emotional Regulation Scale (Hallion et al., 2018)
Self-compassion | Up to 5 months
  Scores on the Self-compassion scale (Neff, 2003)
Motivation for Reducing Self-harm | Up to 5 months
  Scores on the State Motivation for Reducing Self-harm scale (Robinson et al., 2016)
Mystical Experience | Up to 5 months
  Scores on the Mystical Experience questionnaire (Barrett et al., 2015)
Challenging Psychedelic Experience | Up to 5 months
  Scores on the Challenging Experience questionnaire (Barrett et al., 2016)
Emotional Breakthrough | Up to 5 months
  Scores on the Emotional Breakthrough inventory (EBI; Roseman et al., 2019)
Attrition | Up to 5 months
  Percentage of eligible enrolled participants completing outcome assessment

CONTACTS AND LOCATIONS:
Overall Officials: Martina Di Simplicio, Dr, Principal Investigator — Imperial College London; David Nutt, Prof, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All non identifiable outcome measures will be shared.
Supporting Information: Study Protocol
Access Criteria: Data will be publicly available on the OSF repository.

REFERENCES:
- [Background] Passie T, Guss J, Krahenmann R. Lower-dose psycholytic therapy - A neglected approach. Front Psychiatry. 2022 Dec 2;13:1020505. doi: 10.3389/fpsyt.2022.1020505. eCollection 2022. PMID 36532196
- [Background] Doss MK, Povazan M, Rosenberg MD, Sepeda ND, Davis AK, Finan PH, Smith GS, Pekar JJ, Barker PB, Griffiths RR, Barrett FS. Psilocybin therapy increases cognitive and neural flexibility in patients with major depressive disorder. Transl Psychiatry. 2021 Nov 8;11(1):574. doi: 10.1038/s41398-021-01706-y. PMID 34750350
- [Background] Erritzoe D, Roseman L, Nour MM, MacLean K, Kaelen M, Nutt DJ, Carhart-Harris RL. Effects of psilocybin therapy on personality structure. Acta Psychiatr Scand. 2018 Nov;138(5):368-378. doi: 10.1111/acps.12904. Epub 2018 Jun 19. PMID 29923178
- [Background] Roseman L, Demetriou L, Wall MB, Nutt DJ, Carhart-Harris RL. Increased amygdala responses to emotional faces after psilocybin for treatment-resistant depression. Neuropharmacology. 2018 Nov;142:263-269. doi: 10.1016/j.neuropharm.2017.12.041. Epub 2017 Dec 27. PMID 29288686
- [Background] Goodwin GM, Aaronson ST, Alvarez O, Arden PC, Baker A, Bennett JC, Bird C, Blom RE, Brennan C, Brusch D, Burke L, Campbell-Coker K, Carhart-Harris R, Cattell J, Daniel A, DeBattista C, Dunlop BW, Eisen K, Feifel D, Forbes M, Haumann HM, Hellerstein DJ, Hoppe AI, Husain MI, Jelen LA, Kamphuis J, Kawasaki J, Kelly JR, Key RE, Kishon R, Knatz Peck S, Knight G, Koolen MHB, Lean M, Licht RW, Maples-Keller JL, Mars J, Marwood L, McElhiney MC, Miller TL, Mirow A, Mistry S, Mletzko-Crowe T, Modlin LN, Nielsen RE, Nielson EM, Offerhaus SR, O'Keane V, Palenicek T, Printz D, Rademaker MC, van Reemst A, Reinholdt F, Repantis D, Rucker J, Rudow S, Ruffell S, Rush AJ, Schoevers RA, Seynaeve M, Shao S, Soares JC, Somers M, Stansfield SC, Sterling D, Strockis A, Tsai J, Visser L, Wahba M, Williams S, Young AH, Ywema P, Zisook S, Malievskaia E. Single-Dose Psilocybin for a Treatment-Resistant Episode of Major Depression. N Engl J Med. 2022 Nov 3;387(18):1637-1648. doi: 10.1056/NEJMoa2206443. PMID 36322843
- [Background] Holmes EA, Arntz A, Smucker MR. Imagery rescripting in cognitive behaviour therapy: images, treatment techniques and outcomes. J Behav Ther Exp Psychiatry. 2007 Dec;38(4):297-305. doi: 10.1016/j.jbtep.2007.10.007. Epub 2007 Oct 26. PMID 18035331
- [Background] Hasking PA, Di Simplicio M, McEvoy PM, Rees CS. Emotional cascade theory and non-suicidal self-injury: the importance of imagery and positive affect. Cogn Emot. 2018 Aug;32(5):941-952. doi: 10.1080/02699931.2017.1368456. Epub 2017 Aug 25. PMID 28838289
- [Background] Di Simplicio M, Appiah-Kusi E, Wilkinson P, Watson P, Meiser-Stedman C, Kavanagh DJ, Holmes EA. Imaginator: A Proof-of-Concept Feasibility Trial of a Brief Imagery-Based Psychological Intervention for Young People Who Self-Harm. Suicide Life Threat Behav. 2020 Jun;50(3):724-740. doi: 10.1111/sltb.12620. Epub 2020 Feb 14. PMID 32057131
- [Background] Ji JL, Kavanagh DJ, Holmes EA, MacLeod C, Di Simplicio M. Mental imagery in psychiatry: conceptual & clinical implications. CNS Spectr. 2019 Feb;24(1):114-126. doi: 10.1017/S1092852918001487. Epub 2019 Jan 28. PMID 30688194

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT06798636/Prot_SAP_000.pdf